CLINICAL TRIAL: NCT04956250
Title: Traffic Safety Study at Calgary Elementary Schools
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were intended to be directly recruited.
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REB19-1455
Record Dates: First submitted 2021-04-07; First posted 2021-07-09 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2021-03

CONDITIONS: Motor Vehicle Injury

STUDY DESIGN:
Intervention Model Description: Modified Stepped-Wedge Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traffic Calming Curb Group (Experimental): Traffic calming curbs are yellow concrete slabs designed by the City of Calgary to be the same height as other roadside curbs and improve safety by reducing the street width, similar to curb extensions.
  Interventions: Other: Traffic Calming Curbs
- In-Street Sign Group (Experimental): In-street pedestrian signs are regulatory signs placed along the centre line of the street, to remind road users of a pedestrian right-of-way at the marked/unmarked crosswalk.
  Interventions: Other: In-Street Pedestrian Sign

INTERVENTIONS:
Other: Traffic Calming Curbs — Temporary curb extensions, placed at intersections.
  Arms: Traffic Calming Curb Group
Other: In-Street Pedestrian Sign — Yield sign placed in middle of road at intersection.
  Arms: In-Street Sign Group

SUMMARY:
Installing specific traffic calming features designed to reduce vehicle speed and volume around schools may lead to a reduction in injury risk for child pedestrians and bicyclists, and may increase numbers of children walking and bicycling to school. Therefore, this study seeks to evaluate the effectiveness of specific built environment features at influencing traffic speed and volume, and active transportation, both immediately following installation and months later.

DETAILED DESCRIPTION:
Background Collisions with motor-vehicles are a leading cause of severe child bicyclist and pedestrian injuries in Canada. Injury rates and severity are associated with traffic speeds and volume but may be moderated through traffic calming.

Objective To assess the association of specific traffic calming measures on changes in traffic speed and volume, and active transportation prevalence, around Calgary, Alberta, Canada elementary schools.

Design This modified stepped-wedge randomized controlled trial was conducted at a sample of public elementary schools, from July 2020 to May 2021. Schools had either traffic calming curbs or in-street signs installed at an intersection within 100 m of the main entrance. The primary outcome was speed of vehicles driving towards or away from intervention. Secondary outcomes were traffic volume driving past the intervention and counts of children using active transportation at the intervention crosswalk.

ELIGIBILITY:
Inclusion Criteria:

* No individual participants are recruited.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Traffic Speed - Pre-intervention | At each location, a week of pre-intervention data collection will occur a week prior to the intervention being installed.
  Traffic speed of all vehicles who pass by the intervention will be recorded.
Traffic Speed - Post-intervention | At each location, a week of post-intervention data collection will occur a week after the intervention being installed.
  Traffic speed of all vehicles who pass by the intervention will be recorded.
Traffic Speed - Follow-up | At a random selection of locations (drawn from those that received the intervention during the school year), a week of data collection will occur during the spring following the installation of the intervention.
  Traffic speed of all vehicles who pass by the intervention will be recorded.

SECONDARY OUTCOMES:
Traffic Volume - Pre-intervention | At each location, a week of pre-intervention data collection will occur a week prior to the intervention being installed.
  The number of all vehicles who pass by the intervention will be recorded.
Traffic Volume - Post-intervention | At each location, a week of post-intervention data collection will occur a week after the intervention being installed.
  The number of all vehicles who pass by the intervention will be recorded.
Traffic Volume - Follow-up | At a random selection of locations (drawn from those that received the intervention during the school year), a week of data collection will occur during the spring following the installation of the intervention.
  The number of all vehicles who pass by the intervention will be recorded.
Active Transportation Counts - Pre-intervention | At each location, a day of pre-intervention data collection will occur a week prior to the intervention being installed. .
  The number of people (Adults v Children) who use the intervention location, and mode of travel (e.g. walking, bicycling).
Active Transportation Counts - Post-intervention | At each location, a day of post-intervention data collection will occur a week after the intervention being installed. .
  The number of people (Adults v Children) who use the intervention location, and mode of travel (e.g. walking, bicycling).
Active Transportation Counts - Follow-up | At a random selection of locations (drawn from those that received the intervention during the school year), a day of data collection will occur during the spring following the installation of the intervention.
  The number of people (Adults v Children) who use the intervention location, and mode of travel (e.g. walking, bicycling).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada